CLINICAL TRIAL: NCT06562322
Title: Acute Dose-response Effect of Photobiomodulation Therapy on Muscle Performance in Female Futsal Players: a Randomized, Double-blind, Placebo-controlled, Crossover Study
Brief Title: Acute Effect of Photobiomodulation Therapy on Muscle Performance in Female Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Andreo Fernando Aguiar, Principal investigator, Universidade Norte do Paraná
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Photobiomodulation and futsal
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2024-08

CONDITIONS: Muscle Performance; Photobiomodulation Therapy
Keywords: Physical test; Photobiomodulation therapy; Futsal; Light-emitting diodes; Muscle power; Muscle strength

STUDY DESIGN:
Intervention Model Description: Crossover
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo PBMT (Placebo Comparator): Participants will be received placebo PBMT immediately before physical tests.
  Interventions: Device: Placebo
- 300 J PBMT (Active Comparator): Participants will be received PBMT at 300 J immediately before physical tests.
  Interventions: Device: 300 J
- 600 J PBMT (Active Comparator): Participants will be received PBMT at 600 J immediately before physical tests.
  Interventions: Device: 600 J
- 1260 J PBMT (Active Comparator): Participants will be received PBMT at 1260 J immediately before physical tests.
  Interventions: Device: 1260 J

INTERVENTIONS:
Device: Placebo — Participants will be received placebo PBMT on the quadriceps muscle of both legs, immediately before physical tests, using a device containing 200 LEDs (100 red and 100 infrared)
  Arms: placebo PBMT
Device: 300 J — Participants will be received PBMT at 300 J on the quadriceps muscle of both legs, immediately before physical tests, using a device containing 200 LEDs (100 red and 100 infrared)
  Arms: 300 J PBMT
Device: 600 J — Participants will be received PBMT at 600 J on the quadriceps muscle of both legs, immediately before physical tests, using a device containing 200 LEDs (100 red and 100 infrared)
  Arms: 600 J PBMT
Device: 1260 J — Participants will be received PBMT at 1260 J on the quadriceps muscle of both legs, immediately before physical tests, using a device containing 200 LEDs (100 red and 100 infrared)
  Arms: 1260 J PBMT

SUMMARY:
Photobiomodulation therapy (PBMT) has recently been indicated as a potential therapeutic strategy in diverse health and sports contexts. However, its efficacy on muscle performance in female futsal players remains unknown. The purpose of this study was to investigate the dose-response effect of PBMT on muscle performance in female futsal players.

DETAILED DESCRIPTION:
Background: Photobiomodulation therapy (PBMT) has recently been indicated as a potential therapeutic strategy in diverse health and sports contexts. However, its efficacy on muscle performance in female futsal players remains unknown. The purpose of this study is to investigate the dose-response effect of PBMT on muscle performance in female futsal players. Methods: In a crossover design, fifteen female futsal athletes (age: 18-30 years) will be randomized to receive 1 of 4 PBMT conditions (placebo, 300, 900, and 1260 joules [J]) on four occasions, separated by a 2-wk washout period. PBMT treatments will be applied on the quadriceps muscle of both legs using a device containing 200 light-emitting diodes (LEDs), immediately before the following tests (dependent variables): countermovement jump (CMJ) (i.e., flight time as indicator of muscle power), maximum voluntary isometric contraction (MVIC) for the leg extension exercise (i.e., muscle strength), and 3 sets of repetitions-to-failure (i.e., local muscular endurance) for the 45º leg press exercise, with recording of rating of perceived exertion (RPE) after each set. The fatigue index will be determined by the number of repetitions between sets 1 and 3. Statistical analyses will be performe using IBM SPSS Statistics for Windows (version 24.0; IBM Corp., Armonk, NY). Data will be tested for normality and homogeneity using the Shapiro-Wilk's and Levene's tests, respectively. One-way ANOVA tests will be performed to evaluate the differences in the fatigue index, flight time, and peak and mean torque between the treatment conditions (placebo, 300, 900, and 1260 J). Changes over time and between treatment conditions in maximum number of repetitions and RPE will be analyzed with two-way repeated measures ANOVA. Violation of sphericity was corrected using the Greenhouse-Geisser method. When significant differences will be confirmed with the ANOVA, multiple comparison testing will be performed using the Bonferroni post hoc correction to identify these differences. Values will be expressed as mean (standard deviation and 95% confidence interval). The significance level was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years
* Playing futsal regularly for more than 1 year.

Exclusion Criteria:

* Use of any ergogenic or anabolic supplement within 6 months prior to the start of the study,
* Take any medication that may affect the ability to perform the physical tests,
* Have any physical limitation (e.g. joint or muscle injury) that may affect the ability to perform the physical test,
* Be engaged in a restricted diet program (e.g. weight loss diet),
* Have any skin sensitivity or diseases (e.g. erysipelas, eczema, dermatitis, psoriasis and urticaria) in the irradiated area that may be aggravated by PBMT.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Repetitions-to-failure | 10 minutes
  The repetitions-to-failure test in the 45º leg press exercise consists of 3 sets at 70% of 1RM, with a 60-s rest interval between each set. Participants will perform as many repetitions as possible until momentary failure (i.e., when the participant is unable to complete the concentric portion of their current repetition across the full range of motion despite using maximal effort), and the maximum number of repetitions in each set will be recorded.
Fatigue index (FI) | 10 minutes
  The fatigue index (FI) will be determined by the equation: [(REPS3 - REPS1)/REPS1]*100, where: REPS3 = number of repetitions in set 3, multiplied by the load lifted, and REPS1 = number of repetitions in set 1, multiplied by the load lifted. The higher the FI value (%), the higher the level of muscle fatigue.
Rating of perceive exterion (RPE) | 10 minutes
  Rating of perceived exertion (RPE) will be recorded immediately after completion of each set using the OMNI-RES scale. The participants will be instructed to report the perceived exertion value by indicating a number on the OMNI-RES scale (0 for ''no effort'' and 10 for ''maximal effort'') that best represented their momentary exertion.
Countermovement vertical jump (CMJ) | 10 minutes
  The CMJ test will be performed on a force platform (BIOMEC400-412, EMG System to Brazil Ltda, São Paulo, Brazil) to assess the flight time. Participants will perform three CMJs, interspersed with 1 min of rest, and the highest flight time will be used as an indicator of muscle power. The test will began with the participant standing, knees extended, and hands fixed on the iliac crest region (hips). The participant then will flexed their legs at an angle of approximately 90º and then quickly extended their legs to maximize the height of the jump. Hands will be kepted on hips throughout the jump.
Maximum voluntary isometric contraction (MVIC) | 10 minutes
  The MVIC test for the leg extension exercise (bilateral) will be performed using an isometric dynamometer (CEFISE Biotechnology, São Carlos, Brazil). Briefly, participants will perform three MVICs at 120º of knee flexion (180º = full extension) lasting 5 s, interspersed with 5 s of rest. Participants will be instructed and verbally encouraged to exert maximum force during all attempts. The highest value obtained for peak and mean torque of the three MVICs will be used for the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Norte do Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steele J, Fisher J, Giessing J, Gentil P. Clarity in reporting terminology and definitions of set endpoints in resistance training. Muscle Nerve. 2017 Sep;56(3):368-374. doi: 10.1002/mus.25557. Epub 2017 Apr 1. PMID 28044366
- [Background] Robertson RJ, Goss FL, Rutkowski J, Lenz B, Dixon C, Timmer J, Frazee K, Dube J, Andreacci J. Concurrent validation of the OMNI perceived exertion scale for resistance exercise. Med Sci Sports Exerc. 2003 Feb;35(2):333-41. doi: 10.1249/01.MSS.0000048831.15016.2A. PMID 12569225
- [Background] Luque MZ, Aguiar AF, da Silva-Araujo AK, Zaninelli TH, Heintz OK, Saraiva-Santos T, Bertozzi MM, Souza NA, Junior EO, Verri WA Jr, Borghi SM. Evaluation of a preemptive intervention regimen with hesperidin methyl chalcone in delayed-onset muscle soreness in young adults: a randomized, double-blinded, and placebo-controlled trial study. Eur J Appl Physiol. 2023 Sep;123(9):1949-1964. doi: 10.1007/s00421-023-05207-2. Epub 2023 Apr 29. PMID 37119360